CLINICAL TRIAL: NCT03742622
Title: Does Energy Replacement Modify Post-exercise Energy Intake in Adolescents With Obesity?
Brief Title: Energy Intake, Exercise and Energy Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Tza Nou - Maison médicale pour enfants et adolescentes - 230, rue Vercingétorix - B.P. 77 - 63150 La Bourboule (Unknown); SSR Nutrition-Obésité - 33-35 rue Maréchal Leclerc - 63000 Clermont-Ferrand (Unknown); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-415
Record Dates: First submitted 2018-11-06; First posted 2018-11-15 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Pediatric Obesity
Keywords: appetite control; obesity; Adolescents; exercise; Energy replacement
MeSH Terms: conditions — Pediatric Obesity; Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Masking Description: no masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese adolescents (Experimental): 18 adolescents with obesity are involved and will perform the three conditions
  Interventions: Behavioral: CON . control condition without exercise / rest condition; Behavioral: EX. Condition with an acute exercise set in the middle of the morning; Behavioral: EX+R. condition with an acute exercise set in the morning and followed by a energy replacement snack

INTERVENTIONS:
Behavioral: CON . control condition without exercise / rest condition — CON . Control condition without exercise / rest condition. The adolescents will be asked to remain quiet and at rest during the morning and will receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.
Behavioral: EX. Condition with an acute exercise set in the middle of the morning — EX. Condition with an acute exercise set in the middle of the morning The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling) in the morning and will receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals
Behavioral: EX+R. condition with an acute exercise set in the morning and followed by a energy replacement snack — EX+R. condition with an acute exercise set in the morning and followed by a energy replacement snack The adolescents will be asked to complete a 30 minutes exercise set at 65% of their capacities (cycling) in the morning followed by a snack that will cover the whole exercise-induced energy expenditure. They will then receive an ad libitum meal at lunch and dinner times. Their food reward will be assessed before and after lunch. Their appetite feelings will be assessed at regular intervals.

SUMMARY:
The aim of the present study is to compare the effect of an exercise alone versus. An exercise followed by the ingestion of an energy replacement snack on the following energy intake, food reward and appetite feelings in adolescents with obesity.

DETAILED DESCRIPTION:
The present study will compare the nutritional response to the realisation of an acute exercise with and without an energy replacement snack on the following energy intake in adolescents with obesity. 18 adolescents with obesity will be asked to randomly complete three experimental sessions: i) one control session (rest); ii) one session with an acute exercise realized during the morning; iii) one session with the same exercise followed by a snack covering the exercise-induced energy expenditure. Their ad libitum energy intake will be assessed at the following meal as well as at dinner time. Appetite feelings will be assessed at regular intervals and their food reward in response to the lunch will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

* Previous surgical interventions that is considered as non-compatible with the study.
* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-11-17 (Actual); Primary Completion 2019-03-03 (Actual); Study Completion 2019-03-03 (Actual)

PRIMARY OUTCOMES:
Energy intake measured during an ad libitum buffet meal (in kcal). | at lunch (at day 1)
  food intake will be measured ad libitum during a lunch buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using Bilnuts software

SECONDARY OUTCOMES:
Measurement of hunger feelings | at day 1
  hunger area under the curve will be assessed using visual analogue scale through a the day (Leeds Food Preference Questionnaire; LFPQ) Briefly, the LFPQ provides measures of the wanting and liking for an array of food images, varying in both fat content and taste
Food reward | at day 1
  The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ) (Finlayson, King et al. 2008).Briefly, the LFPQ provides measures of the wanting and liking for an array of food images, varying in both fat content and taste

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518